CLINICAL TRIAL: NCT02309801
Title: Human Pharmacology Study to Evaluate the Interaction Between a Natural Inhibitor of Aldehyde Dehydrogenase 2 (ALDH2) and Alcohol in Healthy Volunteers. Pilot Clinical Trial
Brief Title: Interaction Between a Natural Aldehyde Dehydrogenase 2 (ALDH2) Inhibitor and Alcohol
Acronym: COCADEP/2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Ministerio de Sanidad, Servicios Sociales e Igualdad (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: PSMAR/IMIM/COCADEP/2
Record Dates: First submitted 2014-12-03; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — daidzin; Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daidzin and alcohol (Experimental): Daidzin 80 mg, single dose, oral administration (4 capsules of Super-Absorbable Soy Isoflavones®).
  Alcohol 0.5 g/kg (vodka diluted in lemon-flavoured water), single dose, oral administration. Solution of 150 ml.
  Interventions: Dietary Supplement: Daidzin; Dietary Supplement: Alcohol
- Alcohol (Active Comparator): Alcohol 0.5 g/kg (vodka diluted in lemon-flavoured water), single dose, oral administration. Solution of 150 ml.
  Interventions: Dietary Supplement: Alcohol

INTERVENTIONS:
Dietary Supplement: Daidzin — Super-Absorbable Soy Isoflavones, LifeExtension, USA. Single oral dose of 4 capsules (containing 80 mg of daidzin-daidzein).
  Arms: Daidzin and alcohol
Dietary Supplement: Alcohol — Alcohol single oral dose

SUMMARY:
The main objective is to assess whether a natural inhibitor of aldehyde dehydrogenase 2 (ALDH2) contained in a soy extract could interfere on alcohol metabolism and effects in humans.

DETAILED DESCRIPTION:
Soybeans contain isoflavones, which are biologically active polyphenols known as antioxidants and phytoestrogens. These isoflavones include daidzin, daidzein, genistin and glycitin, and have been implicated in the beneficial effects of soy consumption.

Daidzin and daidzein are isoflavones contained in soybean that can act as natural inhibitors of aldehyde dehydrogenase 2. Animal studies have demonstrated that some soy isoflavones can reduce the auto-administration of cocaine and suggest they might be useful to treat cocaine dependence.

Aldehyde dehydrogenase inhibitors, as disulfiram, are currently used in humans to treat alcohol dependence because they interfere with ethanol metabolism (specifically in the transformation of acetaldehyde to acetate.

Alcohol intake after disulfiram administration increases concentration of acetaldehyde in the blood (five to 10 times higher than that found during metabolism of the same amount of alcohol alone). The combination produced acute symptoms of a severe "hangover" (named disulfiram-like reaction), and the patient may experience symptoms as flushing of the skin, tachycardia, shortness of breath, nausea, vomiting, throbbing headache, visual disturbances, mental confusion, and in some cases severe reactions as postural syncope, and circulatory collapse.

In addition, disulfiram have demonstrated clinical efficacy in cocaine dependence. The mechanism of action for that effects are related to its ability to decrease dopamine degradation by inhibiting the dopamine-beta-hydroxylase enzyme (metabolizes dopamine to norepinephrine), and increasing its concentrations in some areas of the brain.

The aim of the study is to assess whether a soy extract containing isoflavones (daidzin, daidzein and genistein) could interfere on alcohol metabolism and produce adverse effects in humans.

ELIGIBILITY:
Inclusion Criteria:

* Understanding and accepting the study procedures and signing the informed consent
* Clinical history and physical examination demonstrating no organic or psychiatric disorders
* The ECG and general blood and urine laboratory tests performed before the study should be within normal ranges. Minor or occasional changes from normal ranges are accepted if, in the investigator's opinion, considering the current state of the art, they are not clinically significant, are not life-threatening for the subjects and do not interfere with the product assessment. These changes and their non-relevance will be justified in writing specifically
* The body mass index (BMI=weigh/height2) will range from 19 to 27 kg/m2, and the weight from 50 to 100 kg
* Ethanol consumption of minimum 2 units per week and previous experience with ethanol intoxication
* Women with regular menstrual cycle (26-32 days)

Exclusion Criteria:

* Not meeting the inclusion criteria
* History or clinical evidence of alcoholism, psychiatric disorders, drug abuse or dependence, or regular use of psychoactive drugs
* Having suffered any organic disease or major surgery in the three months prior to the study start
* Smokers
* Consumption of more than five coffees, teas, colas, other stimulant or xanthine beverages daily in the three months prior to the beginning of the study
* Taking more than 20 g of alcohol per day in women and 40 g of alcohol per day in men
* Regular use of any drug in the month prior to the study sessions.The treatment with single or limited doses of symptomatic medicinal products in the week prior to the study sessions will not be a reason for exclusion if it is calculated that it has been cleared completely the day of the experimental session
* Blood donation 8 weeks before or participation in other clinical trials with drugs in the previous 12 weeks
* Subjects with allergy, intolerance or adverse reactions to alcohol, soya and lactose.
* History or clinical evidence of gastrointestinal, liver, renal or other disorders which may lead to suspecting a disorder in drug absorption, distribution, metabolism or excretion, or that suggest gastrointestinal irritation due to drugs
* Subjects unable to understand the nature, consequences of the study and the procedures requested to be followed
* Subjects with positive serology to Hepatitis B, C or HIV
* Pregnant or breastfeeding women. Women not using effective contraceptive methods
* History or presence of breast cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time curve (AUC 2-10h) | From 2h to 10h after the first administration
  Calculation of AUC for blood alcohol concentrations

SECONDARY OUTCOMES:
Change in signs and symptoms of disulfiram-like reaction | From baseline to 10h after the first administration
  Vital signs (heart rate, blood pressure, respiration rate, oral and facial temperature) and adverse effects measured by visual analogue scales (nausea, vomiting, vertigo, dizziness, headache, breathing difficulty, facial flushing)
Change in drunkenness and euphoria effects | From baseline to 10h after the first administration
  Drunkenness and euphoria will be measured by a visual analogue scale (VAS).
Area Under the Concentration-Time curve (AUC 0-10h) | From baseline to 24h after the first administration
  Calculation of AUC of plasmatic concentrations of daidzein, genistein and equol
Number of participants with Serious and non-serious adverse events | 3 days after each condition
  Collection of adverse events spontaneously reported by the participants and/or observed by the investigators.
Change in other subjective effects | From baseline to 10h after the first administration
  Subjective effects will be measured with the Addiction Research Center Inventory (ARCI)
Elimination half-life | From 2h to 10h after the first administration
  Calculation of elimination half-life from blood ethanol concentrations
Elimination half-life | From baseline to 24h after the first administration
  Calculation of elimination half-life of plasmatic concentrations of daidzein, genistein and equol
Cumulative amount of drug excreted into urine up to collection time | From baseline to 24h after the first administration
  Urine will be collected in the following periods:0-2h,2-8h,8-14h,14-24 h after administration. Concentrations of daidzein, genistein and equol will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Magí Farré, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Parc de Salut Mar., Barcelona, Barcelona, Spain